CLINICAL TRIAL: NCT07259382
Title: Neuro-Inflammation in Extremity Trauma: Risk Verification in Elbow Trauma: The NERVE Pilot Cohort Study
Brief Title: Neuro-Inflammation in Extremity Trauma: Risk Verification in Elbow Trauma: The NERVE Study
Acronym: NERVE
Status: Not yet recruiting | Type: Observational
Sponsor: Université de Montréal (Other)
Responsible Party: Principal Investigator, Dominique Rouleau, Orthopaedic surgeon, Université de Montréal
Other Study IDs: NERVE
Record Dates: First submitted 2025-09-16; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Elbow Dislocation; Elbow Fractures; Inflammation Biomarkers; TBI Traumatic Brain Injury; Nerve Injury
Keywords: Biomarkers; Elbow fracture; elbow dislocation; Nerve injury; TBI
MeSH Terms: conditions — Elbow Fractures; Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Bloodtest
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Elbow fracture: Patient with an acute, isolated elbow fracture
  Interventions: Other: Biomarkers evaluation
- Elbow fracture and peripheral nerve injury: Patient with an acute elbow fracture and a peripheral nerve injury
  Interventions: Other: Biomarkers evaluation
- Ebow fracture and TBI: Patient with an acute elbow fracture and a mild TBI
  Interventions: Other: Biomarkers evaluation

INTERVENTIONS:
Other: Biomarkers evaluation — Participants will undergo blood test that evaluate several inflammatory biomarkers before and after the surgery

SUMMARY:
The primary goal of this proposal is to improve the understanding of the mechanisms causing persistent pain and disability in elbow fracture patients and their associated functional limitations. The specific objectives are as follows for elbow fractures:

1) To describe NI mechanisms using biomarkers; 2) To identify factors related to increased NI biomarkers level; 3) To describe the associations between NI and outcomes; 4) To use these findings to refine a larger fully powered prognostic cohort study Hypotheses

1. Level of neuro-inflammation (NI) biomarkers* will be significantly higher in patients presenting with both elbow fracture and CNS injury or PNI.
2. Consumption of opioid in mg of morphine equivalent will be higher in patients with a higher level of NI biomarkers.
3. Function, assessed by validated joint and limb specific functional questionnaires and QoL will be worse in patients with a higher level of NI biomarkers.
4. Chronic pain at 3 months will be higher (McGill Pain questionnaire V2, Neuropathic pain questionnaire, NPRS) in patients with a higher level of NI biomarkers.
5. Duration of tourniquet use and nerve dissection will be correlated to elbow fracture outcome with a higher level of NI biomarkers.

   * Target biomarkers based on preliminary study will include, but not be limited to: TNFa, IL6, Substance P, IL-1B, TREM-2, IL-16, CCL22, VEGF-a, BMPs (table 1).

DETAILED DESCRIPTION:
Chronic pain after limb fractures remains a challenging clinical problem although scientific and technological advances have made major contributions to improve patient outcomes. Nonetheless, even with an anatomical restoration of the bone architecture, many patients still have major functional limitations and persistent pain. This results in a work productivity loss. In the United States, upper limb injuries generate the highest direct and indirect costs (740M$), followed by lower limb fractures (562M$). Although outcomes following a fracture vary significantly, a "simple" fracture occurring at any time can become a turning point in the patient's life, where they can no longer achieve their pre-fracture functional status. The Canadian Pain Task Force estimates that 8 million Canadians suffer from chronic pain, costing $40 billion annually. This includes a large and understudied group of patients with post traumatic chronic pain, which occurs in up to 50% of patients following fractures. For these patients, opioids are meant to alleviate pain, but substance use disorder is a common problem. Indeed, approximately half of all patients with fractures have significant pain leading to persistent opioid intake 3 months post injury and 40% will suffer from a neuropathic type of pain, which is poorly controlled by medications. Opioid use is also associated with an increased sensitivity to pain (hyperalgesia) and patient dissatisfaction with injury outcome. Complications from prolonged opioid use are numerous, varying from constipation to overdose death. Canada is second worldwide, behind the United States, when it comes to opioid use and mortality. The majority of opioid dependant users were first exposed to opioids through medical prescriptions. This makes it imperative to improve the understanding of pain mechanisms to find alternative treatments to opioids in the management of these injuries.

In clinical practice, it is striking to see how two patients with a similar injury can exhibit completely opposite outcomes: one who has completely healed from the injury and the other with a stiff and painful joint. The reasons for these variations are unclear. A study have shown that only 3.3% of the differences in patient pain levels could be attributed to fracture severity. Given the enormous societal burden of limb injuries it is time for research to investigate the factors that contribute to the 97% of unexplained variability related to post fracture pain. The investigator working hypothesis is that the variability in post-fracture pain is caused by differences in expression of specific proinflammatory cytokines with nociceptive effects. This would explain why most studies strictly focusing on the orthopedic component of limb injury have yielded little improvement in preventing the adverse outcomes experienced by patients, namely chronic pain and loss of function.

Basic science studies have shown that in chronic pain cases, the resolution process following initial inflammation is deficient, leading to an excessive inflammatory response spreading throughout the nervous system long after the injury. This response, globally referred to as neuroinflammation (NI), has been associated with central sensitization, central nervous system (CNS) hyperactivity, allodynia and hyperalgesia. Surprisingly, NI is hardly studied in acute fracture cases, which is shocking given that it could explain chronic pain and disability. Also, some surgical factors may increase peripheral nerve injury (PNI).

Among all upper limb fractures, elbow trauma is the injury most frequently associated with a severe impact on patient function and quality of life. One of the main causes for poor outcomes is the complexity of the elbow joint, which involves three bones and two planes of motion, essential to the position of the hand in space. The flexion extension axis is crucial for eating and hygiene, while forearm pro-supination is mandatory for most professions, from office work to manual labour. Following surgical treatment of an elbow fracture, patients often present with complications, even with adequate bone healing. Indeed, one third of patients complain of ulnar nerve symptoms after distal humerus fracture fixation, and 50% of patients treated surgically for elbow fracture-dislocations will have disabling stiffness and chronic pain. The elbow is ideal to study neuroinflammation and pain as it involves 3 major nerves close to the joint: the radial, ulnar and median nerves. Elbow injury also has a high incidence of associated mild traumatic brain injury (MTBI) and peripheral nerve injury (PNI), 20% and 15% respectively.

1.2 Neuroinflammation Neuroinflammation (NI) can take different forms: central and peripheral. Prevouis investigator's results showed that 23.5% of isolated limb injuries also exhibit a mild traumatic brain injury (mTBI). More specifically, the investigators reported that 20% of ambulatory patients with an elbow fracture have a traumatic brain injury (TBI). Previous studies done by the investigator's team showed that outcomes of patients with a TBI, even mTBI, and a fracture is much poorer, compared to a group of similar patients without TBI, causing a work cessation three time longer (averaging 299 days versus 105 days). Central NI alters acute pain and increases the risk of chronic pain following a limb injury. At the time of brain trauma, brain-resident cells, such as microglia, will produce cytokines and other inflammatory mediators that spread through the peripheral circulatory system causing hypersensitivity and peripheral pain. Damage to the blood-brain barrier (BBB) following traumatic injury, allows circulating peripheral immune cells, produced in response to the fracture and present in high numbers at the site of injury and in immune organs, and the released cytokines to reach the brain and create a hyperactive inflammatory state. Astrocytes and endothelial cells also play a key role in this phenomenon. Importantly, research on US military veterans with orthopaedic injuries has revealed that the presence of mTBI significantly increases the risk of chronic pain and NI, as measured by higher levels of TNF and IL-6. A recent article in Nature also reported that the combined impact of mTBI and fracture to the brain could be permanent, because of the brain's immune memory. Therefore, both the traumatized brain and the fractured limb will evolve more poorly than if each lesion had occurred independently.

There is a spectrum of PNI that can occur at the time of the fracture or during their surgical treatment. It is estimated that these lesions affect between 3% and 10% of trauma extremity patients. In the elbow, certain types of injuries have a much higher rate of PNI; up to 30%. The most benign are called neuropraxia and consist of segmental demyelination. The symptoms include numbness and weakness for a period ranging from a few days to a few weeks. Axonotmesis is a rupture of the axons while the nerve sheath remains intact. Spontaneous healing is possible but will take months. Severe lesions consist in a complete nerve rupture, called neurotmesis. This is rare and requires surgical treatment. The precise incidence of neuropraxia is unknown, because pain following a trauma often hides neurological injury symptoms that heal on their own. These transient lesions contribute to the chronic pain mechanisms, which often lead to persistent opioid consumption.

Neuroinflammation can be the result of an altered, uncontrolled immune response to the peripheral injury. Proinflammatory cytokines such as TNF, IL-1, and IL-6 are rapidly produced after injury, and sometimes expressed for prolonged periods of time if there is no resolution of inflammation solve. Importantly, these proinflammatory cytokines play a major role in the transition from acute to chronic pain, acting as potent mediators of excitatory activity in the CNS through modulation of the glutaminergic system. This increase in excitatory activity also decreases the gamma-aminobutyric acid (GABA) activity, which further affects CNS homeostasis. Neuroinflammation markers consequently increase in the circulatory system. Preliminary experiments in patients with fractures found a strong correlation between plasma levels of proinflammatory cytokines, as well as some less frequently studied biomarkers such as C1qA, and chronic pain. Notably, the C1qA protein was involved in the development of neuropathic pain in animal models and showed variations related to the sex of rodents. In an ongoing study, the investigators demonstrated that NI biomarkers played a role in pain and outcome after human fracture, including TREM2, IL16, CCL22, VEGF-a (appendix), amongst others.

1.3 Surgical factors A literature review shows that tourniquet use and nerve dissection may play a role in elbow surgery outcome. While a tourniquet is often used to avoid bleeding and give better visibility, the tourniquet causes an inflammatory ischemia/reperfusion reaction. Several studies have shown an impact of the tourniquet on pain in lower limb surgery. Using a tourniquet to treat ankle fractures is associated with a greater consumption of opioids for the first 24 hours and more pain at 5 days and 6 weeks post-surgery. Tourniquet duration was also correlated with increased opioid consumption in a Danish study on 603 patients; patients took 0,43 mg more morphine for each additional 10 minutes with the tourniquet. Furthermore, British Medical Council Neurology guidelines for tourniquet use report an increased risk of complex regional pain syndrome in surgeries with a tourniquet. Peripheral nerve ischemia during tourniquet use, for up to 120 minutes, could promote NI. However, there is a lack of data specific to elbow surgery and tourniquet use, as reported by a meta-analysis. Surgical nerve dissection may also cause peripheral nerve inflammation. A recent systematic review of elbow fractures reported that ulnar nerve transposition is related to more chronic symptoms than nerve identification only. The quality of the articles involved in the review was modest and electromyography (EMG) was not used to measure impairment.

In summary, limb fractures are associated with a high risk of sequelae, even with proper healing of osseous and ligamentous components. Pain and disability leading to chronic opioid intake is a major concern. Elbow joint fractures are an excellent subgroup to study this phenomenon because of the high incidence of concomitant central and peripheral neurological injuries. Moreover, having a homogenous patient group will make it easier to compare functional outcomes with joint specific questionnaires and functional evaluation. The Nerve pilot study is well supported by the basic science literature and designed to study the mechanisms leading to neuro-inflammation in injured human patients, with the long-term goal of understanding factors increasing NI (e.g., concomitant head injury, peripheral nerve injury, surgical factors, demographic characteristics) and its consequences (e.g., acute and chronic pain, disability). It is expected that studying the surgical factors that increase NI will allow surgeons to choose different therapeutic options.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years or older with an acute elbow fracture and/or dislocation less than a week old
* Open surgery as the chosen treatment

Exclusion Criteria:

* Patient with a history of ipsilateral upper limb trauma or pathology, neurological disorder.
* Patient unable to answer questionnaires.
* Patient unavailable for a one-year follow-up, for example from another country.
* Patient with vascular injury or open fracture
* Patient with an active inflammatory disease (ex: rheumatoid arthritis)
* Patient using anti-inflammatory drugs or immunosuppressants at the time of the injury.
* Patient with another acute ipsilateral injury to the upper limb
* Polytrauma patients with other injuries than the elbow fracture and concomitant central or peripheral neurological injury.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with an acute elbow surgery with an appointment at the Hôpital du Sacré-Coeur de Montréal
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Biomarkers | Baseline, preoperative, perioperative, immediatly after the intervention, 3months
  Five blood samples per subject will be taken at selected intervals to measure the serum levels of the targeted pro-inflammatory cytokines for the 60 selected patients. A blood sample will be collected at the first appointment before surgery. Preoperative and postoperative blood samples will also be collected in the operating room. The first will be taken before skin asepsis and the second will be taken immediately after application of the final wound dressing. Blood from the fracture site (hematoma) will also be collected when possible. The fifth blood sample will be collected at 3 months of follow up. Samples will be stored in a -70°C freezer in each city and sent every 6 months for analysis to Olink, Montreal. Group dosage will be performed for the NI factors and circulating proteins (e.g. cytokines, chemokines, neuropeptides), such as TNF, IL-1, IL-6, IL-16, osteopontin, S100B, NSE, GFAP, Substance P, TREM-2, CCL22, and BMPs.

SECONDARY OUTCOMES:
PREE | Baseline, preop, 2 weeks, 3-6-12 months
  The PREE is a validated patient-reported outcome measure designed to assess pain and functional limitations related to elbow disorders. It consists of 20 items divided into two subscales:
  Pain Subscale (5 items): Measures pain intensity during various activities. Function Subscale (15 items): Assesses difficulty in performing specific and usual daily activities.
  Each item is rated on a scale from 0 (no pain or difficulty) to 10 (worst pain or complete inability). A total score out of 100 is calculated by combining both subscales with equal weighting. Higher scores indicate greater pain and disability.
  Method of Measurement: Self-administered questionnaire completed by participants.
Range of motion | Baseline, preop, immediatly after the procedure, 2 weeks, 3-6-12months
  Participant will undergo a range of motion evaluation of the elbow at each time frame, if possible. ROM evaluation will include flexion, extension, pronation and supination. Evaluation will be done with a numeric goniometer by a physicial therapist and evaluate in degree
Pain assessment | Baseline, preop, 2 weeks, 3-6-12 months
  Visual analog pain scale from 0 to 10. 0 would be no pain, 10 worst pain
Opioïds consumption | Recorded once per day from baseline through 12months
  Daily medication diary
Quick-DASH | Baseline, preop, 2weeks, 3 months, 6 months, 12 months
  Description:
  The QuickDASH is a patient-reported outcome measure used to assess physical function and symptoms in individuals with upper limb disorders. It consists of 11 items rated on a 5-point Likert scale. The total score is transformed to a 0-100 scale, with higher scores indicating greater disability. It is validated for use in clinical trials and is sensitive to changes over time.
  Method of Measurement:
  Self-administered questionnaire completed by participants.
EQ-5D-5L | Baseline, pre-op, 2 weeks, 3-6-12 months
  he EQ-5D-5L is a standardized instrument for measuring health-related quality of life. It includes five dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression), each rated on five levels of severity. It also includes a Visual Analogue Scale (EQ VAS) where participants rate their overall health from 0 to 100. Responses can be converted into a single index value using validated scoring algorithms. Higher index values and VAS scores indicate better health status.
  Method of Measurement:
  Self-administered questionnaire completed by participants.
Rivermead | Baseline, pre-op, 2 weeks, 3-6-12 months
  The RPQ is a patient-reported outcome measure used to assess the severity of post-concussion symptoms following traumatic brain injury. It includes 16 items rated on a 5-point scale, comparing current symptoms to pre-injury status. The questionnaire is divided into two scoring clusters: RPQ-3 (early physical symptoms) and RPQ-13 (later cognitive and emotional symptoms). Total scores range from 0 to 64, with higher scores indicating greater symptom severity. The RPQ is validated and widely used in concussion research and clinical practice
  Method of Measurement:
  Self-administered questionnaire completed by participants.
S-LANSS | Baseline, pre-op, 2 weeks, 3-6-12 months
  The S-LANSS is a self-administered questionnaire used to identify pain of predominantly neuropathic origin. It includes 7 items assessing sensory symptoms and pain characteristics. Each item is scored, and a total score of 12 or more indicates likely neuropathic pain. The tool is validated for use in clinical and postal research and does not require physical examination.
  Method of Measurement:
  Self-administered questionnaire completed by participants.
SF-MPQ | Baseline, pre-op, 2 weeks, 3-6-12 months
  Description:
  The SF-MPQ-2 is a patient-reported outcome measure used to assess the intensity and quality of pain across multiple dimensions. It includes 22 descriptors rated on an 11-point scale (0-10), covering continuous, intermittent, neuropathic, and affective pain. Scores are calculated for each category and as a total score. Higher scores indicate greater pain severity. The SF-MPQ-2 is validated for use in diverse pain populations and is sensitive to treatment-related changes.
  Method of Measurement:
  Self-administered questionnaire completed by participants.
Peripheral nerve injury classification (PNI) | Baseline, preop, immediatly after the procedure, 2 weeks, 3-6-12months
  Clinical evidence of PNI will be determined with an assessment of strength and sensitivity of the 3 nerves (radial (anterior and posterior branches), median, ulnar).
  Allodynia: On the healthy and affected side, the evaluator will apply a series of monofilaments.
  Methodology: the patient will be seated with his eyes closed. We will start by applying the 4.17 monofilament on the healthy side and then increase to the 4.93 monofilament. The patient will have to answer yes or no if he feels pain. We will do the same on the affected side Hypoesthesia: On the healthy side and affected side, the evaluator will apply the following monofilaments: Radial nerve: 3.61,Median nerve: 3.22,Ulnar nerve: 3.22 Methodology: the patient will be seated with his eyes closed. If the patient does not feel pressure from the monofilament, the evaluator continues to increase the monofilament grades until the patient feels pressure.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mahabier KC, Hartog DD, Van Veldhuizen J, Panneman MJ, Polinder S, Verhofstad MH, Van Lieshout EM. Trends in incidence rate, health care consumption, and costs for patients admitted with a humeral fracture in The Netherlands between 1986 and 2012. Injury. 2015 Oct;46(10):1930-7. doi: 10.1016/j.injury.2015.07.025. Epub 2015 Aug 4. PMID 26296455
- [Result] Jodoin M, Rouleau DM, Therrien E, Chauny JM, Sandman E, Larson-Dupuis C, Leduc S, Gosselin N, De Beaumont L. Investigating the incidence and magnitude of heterotopic ossification with and without joints involvement in patients with a limb fracture and mild traumatic brain injury. Bone Rep. 2019 Aug 13;11:100222. doi: 10.1016/j.bonr.2019.100222. eCollection 2019 Dec. PMID 31463337
- [Result] Chapleau J, Canet F, Petit Y, Sandman E, Laflamme GY, Rouleau DM. Demographic and anthropometric factors affecting elbow range of motion in healthy adults. J Shoulder Elbow Surg. 2013 Jan;22(1):88-93. doi: 10.1016/j.jse.2012.05.028. Epub 2012 Sep 1. PMID 22947233
- [Result] Rouleau DM, Sandman E, van Riet R, Galatz LM. Management of fractures of the proximal ulna. J Am Acad Orthop Surg. 2013 Mar;21(3):149-60. doi: 10.5435/JAAOS-21-03-149. PMID 23457065
- [Result] Thabane L, Lancaster G. A guide to the reporting of protocols of pilot and feasibility trials. Pilot Feasibility Stud. 2019 Feb 28;5:37. doi: 10.1186/s40814-019-0423-8. eCollection 2019. PMID 30858987
- [Result] Zetterberg H, Blennow K. Fluid biomarkers for mild traumatic brain injury and related conditions. Nat Rev Neurol. 2016 Oct;12(10):563-74. doi: 10.1038/nrneurol.2016.127. Epub 2016 Sep 16. PMID 27632903
- [Result] Niezgoda A, Michalak S, Losy J, Kalinowska-Lyszczarz A, Kozubski W. sNCAM as a specific marker of peripheral demyelination. Immunol Lett. 2017 May;185:93-97. doi: 10.1016/j.imlet.2017.03.011. Epub 2017 Mar 21. PMID 28336415
- [Result] Oh YM, Ma TZ, Kwak YG, Eun JP. Proteomic evaluation to identify biomarkers for carpal tunnel syndrome: a comparative serum analysis. Connect Tissue Res. 2013;54(1):76-81. doi: 10.3109/03008207.2012.746320. Epub 2012 Dec 3. PMID 23186247
- [Result] Michetti F, D'Ambrosi N, Toesca A, Puglisi MA, Serrano A, Marchese E, Corvino V, Geloso MC. The S100B story: from biomarker to active factor in neural injury. J Neurochem. 2019 Jan;148(2):168-187. doi: 10.1111/jnc.14574. Epub 2018 Nov 12. PMID 30144068
- [Result] Bergquist ER, Hammert WC. Timing and appropriate use of electrodiagnostic studies. Hand Clin. 2013 Aug;29(3):363-70. doi: 10.1016/j.hcl.2013.04.005. Epub 2013 Jun 12. PMID 23895716
- [Result] Seddon HJ. A Classification of Nerve Injuries. Br Med J. 1942 Aug 29;2(4260):237-9. doi: 10.1136/bmj.2.4260.237. No abstract available. PMID 20784403
- [Result] Packham TL, Spicher CJ, MacDermid JC, Quintal I, Buckley N. Evaluating a sensitive issue: reliability of a clinical evaluation for allodynia severity. Somatosens Mot Res. 2020 Mar;37(1):22-27. doi: 10.1080/08990220.2019.1704242. Epub 2019 Dec 20. PMID 31858880
- [Result] Chichery R, Chichery MP. Motor and behavioural effects induced by putative neurotransmitter injection into the optic lobe of the cuttlefish, Sepia officinalis. Comp Biochem Physiol C Comp Pharmacol Toxicol. 1985;80(2):415-9. doi: 10.1016/0742-8413(85)90078-7. PMID 2861029
- [Result] Houdek MT, Shin AY. Management and complications of traumatic peripheral nerve injuries. Hand Clin. 2015 May;31(2):151-63. doi: 10.1016/j.hcl.2015.01.007. Epub 2015 Feb 28. PMID 25934193
- [Result] King NS, Crawford S, Wenden FJ, Moss NE, Wade DT. The Rivermead Post Concussion Symptoms Questionnaire: a measure of symptoms commonly experienced after head injury and its reliability. J Neurol. 1995 Sep;242(9):587-92. doi: 10.1007/BF00868811. PMID 8551320
- [Result] Teasdale G, Jennett B. Assessment of coma and impaired consciousness. A practical scale. Lancet. 1974 Jul 13;2(7872):81-4. doi: 10.1016/s0140-6736(74)91639-0. No abstract available. PMID 4136544
- [Result] Nazari G, MacDermid JC, Bain J, Levis CM, Thoma A. Estimation of health-related-quality of life depends on which utility measure is selected for patients with carpal tunnel syndrome. J Hand Ther. 2017 Jul-Sep;30(3):299-306. doi: 10.1016/j.jht.2016.11.001. Epub 2016 Dec 14. PMID 27988154
- [Result] Cook KF, Dunn W, Griffith JW, Morrison MT, Tanquary J, Sabata D, Victorson D, Carey LM, Macdermid JC, Dudgeon BJ, Gershon RC. Pain assessment using the NIH Toolbox. Neurology. 2013 Mar 12;80(11 Suppl 3):S49-53. doi: 10.1212/WNL.0b013e3182872e80. PMID 23479545
- [Result] Bennett M. The LANSS Pain Scale: the Leeds assessment of neuropathic symptoms and signs. Pain. 2001 May;92(1-2):147-57. doi: 10.1016/s0304-3959(00)00482-6. PMID 11323136
- [Result] Hawker GA, Mian S, Kendzerska T, French M. Measures of adult pain: Visual Analog Scale for Pain (VAS Pain), Numeric Rating Scale for Pain (NRS Pain), McGill Pain Questionnaire (MPQ), Short-Form McGill Pain Questionnaire (SF-MPQ), Chronic Pain Grade Scale (CPGS), Short Form-36 Bodily Pain Scale (SF-36 BPS), and Measure of Intermittent and Constant Osteoarthritis Pain (ICOAP). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S240-52. doi: 10.1002/acr.20543. No abstract available. PMID 22588748
- [Result] Lovejoy TI, Turk DC, Morasco BJ. Evaluation of the psychometric properties of the revised short-form McGill Pain Questionnaire. J Pain. 2012 Dec;13(12):1250-7. doi: 10.1016/j.jpain.2012.09.011. PMID 23182230
- [Result] Fayad F, Lefevre-Colau MM, Gautheron V, Mace Y, Fermanian J, Mayoux-Benhamou A, Roren A, Rannou F, Roby-Brami A, Revel M, Poiraudeau S. Reliability, validity and responsiveness of the French version of the questionnaire Quick Disability of the Arm, Shoulder and Hand in shoulder disorders. Man Ther. 2009 Apr;14(2):206-12. doi: 10.1016/j.math.2008.01.013. Epub 2008 Apr 23. PMID 18436467
- [Result] Beauchemin G, MacDermid JC, Bourduas K, Poirier MF, Gaudelli C, Rouleau DM. Translation and validation of the PREE (Patient Rated Elbow Evaluation) to a French version. Orthop Traumatol Surg Res. 2015 Jun;101(4):405-9. doi: 10.1016/j.otsr.2015.03.012. Epub 2015 Apr 27. PMID 25936242
- [Result] Vincent JI, MacDermid JC, King GJ, Grewal R. Rasch analysis of the Patient Rated Elbow Evaluation questionnaire. Health Qual Life Outcomes. 2015 Jun 20;13:84. doi: 10.1186/s12955-015-0275-8. PMID 26092294
- [Result] de Mos M, Laferriere A, Millecamps M, Pilkington M, Sturkenboom MC, Huygen FJ, Coderre TJ. Role of NFkappaB in an animal model of complex regional pain syndrome-type I (CRPS-I). J Pain. 2009 Nov;10(11):1161-9. doi: 10.1016/j.jpain.2009.04.012. PMID 19878863
- [Result] van der Velde J, Serfontein L, Iohom G. Reducing the potential for tourniquet-associated reperfusion injury. Eur J Emerg Med. 2013 Dec;20(6):391-6. doi: 10.1097/MEJ.0b013e3283591668. PMID 22990037
- [Result] Konrad G, Markmiller M, Lenich A, Mayr E, Ruter A. Tourniquets may increase postoperative swelling and pain after internal fixation of ankle fractures. Clin Orthop Relat Res. 2005 Apr;(433):189-94. doi: 10.1097/01.blo.0000151849.37260.0a. PMID 15805957
- [Result] Kruse H, Christensen KP, Moller AM, Gogenur I. Tourniquet use during ankle surgery leads to increased postoperative opioid use. J Clin Anesth. 2015 Aug;27(5):380-4. doi: 10.1016/j.jclinane.2015.03.034. Epub 2015 May 12. PMID 25979462
- [Result] Shearin JW, Chapman TR, Miller A, Ilyas AM. Ulnar Nerve Management with Distal Humerus Fracture Fixation: A Meta-Analysis. Hand Clin. 2018 Feb;34(1):97-103. doi: 10.1016/j.hcl.2017.09.010. PMID 29169602
- [Result] Stewart AN, Lowe JL, Glaser EP, Mott CA, Shahidehpour RK, McFarlane KE, Bailey WM, Zhang B, Gensel JC. Acute inflammatory profiles differ with sex and age after spinal cord injury. J Neuroinflammation. 2021 May 13;18(1):113. doi: 10.1186/s12974-021-02161-8. PMID 33985529
- [Result] Olivecrona C, Ponzer S, Hamberg P, Blomfeldt R. Lower tourniquet cuff pressure reduces postoperative wound complications after total knee arthroplasty: a randomized controlled study of 164 patients. J Bone Joint Surg Am. 2012 Dec 19;94(24):2216-21. doi: 10.2106/JBJS.K.01492. PMID 23318611
- [Result] Du H, Shi J, Wang M, An S, Guo X, Wang Z. Analyses of gene expression profiles in the rat dorsal horn of the spinal cord using RNA sequencing in chronic constriction injury rats. J Neuroinflammation. 2018 Sep 25;15(1):280. doi: 10.1186/s12974-018-1316-0. PMID 30253787
- [Result] Guo TZ, Wei T, Huang TT, Kingery WS, Clark JD. Oxidative Stress Contributes to Fracture/Cast-Induced Inflammation and Pain in a Rat Model of Complex Regional Pain Syndrome. J Pain. 2018 Oct;19(10):1147-1156. doi: 10.1016/j.jpain.2018.04.006. Epub 2018 Apr 30. PMID 29715519
- [Result] Uceyler N, Eberle T, Rolke R, Birklein F, Sommer C. Differential expression patterns of cytokines in complex regional pain syndrome. Pain. 2007 Nov;132(1-2):195-205. doi: 10.1016/j.pain.2007.07.031. Epub 2007 Sep 24. PMID 17890011
- [Result] Schmid AB, Coppieters MW, Ruitenberg MJ, McLachlan EM. Local and remote immune-mediated inflammation after mild peripheral nerve compression in rats. J Neuropathol Exp Neurol. 2013 Jul;72(7):662-80. doi: 10.1097/NEN.0b013e318298de5b. PMID 23771220
- [Result] Schlereth T, Drummond PD, Birklein F. Inflammation in CRPS: role of the sympathetic supply. Auton Neurosci. 2014 May;182:102-7. doi: 10.1016/j.autneu.2013.12.011. Epub 2013 Dec 22. PMID 24411269
- [Result] Block L. Glial dysfunction and persistent neuropathic postsurgical pain. Scand J Pain. 2016 Jan;10:74-81. doi: 10.1016/j.sjpain.2015.10.002. Epub 2015 Nov 13. PMID 28361776
- [Result] Liu XG, Pang RP, Zhou LJ, Wei XH, Zang Y. Neuropathic Pain: Sensory Nerve Injury or Motor Nerve Injury? Adv Exp Med Biol. 2016;904:59-75. doi: 10.1007/978-94-017-7537-3_5. PMID 26900063
- [Result] Moreau N, Mauborgne A, Bourgoin S, Couraud PO, Romero IA, Weksler BB, Villanueva L, Pohl M, Boucher Y. Early alterations of Hedgehog signaling pathway in vascular endothelial cells after peripheral nerve injury elicit blood-nerve barrier disruption, nerve inflammation, and neuropathic pain development. Pain. 2016 Apr;157(4):827-839. doi: 10.1097/j.pain.0000000000000444. PMID 26655733
- [Result] Martins RS, Bastos D, Siqueira MG, Heise CO, Teixeira MJ. Traumatic injuries of peripheral nerves: a review with emphasis on surgical indication. Arq Neuropsiquiatr. 2013 Oct;71(10):811-4. doi: 10.1590/0004-282X20130127. PMID 24212521
- [Result] Wendeln AC, Degenhardt K, Kaurani L, Gertig M, Ulas T, Jain G, Wagner J, Hasler LM, Wild K, Skodras A, Blank T, Staszewski O, Datta M, Centeno TP, Capece V, Islam MR, Kerimoglu C, Staufenbiel M, Schultze JL, Beyer M, Prinz M, Jucker M, Fischer A, Neher JJ. Innate immune memory in the brain shapes neurological disease hallmarks. Nature. 2018 Apr;556(7701):332-338. doi: 10.1038/s41586-018-0023-4. Epub 2018 Apr 11. PMID 29643512
- [Result] Kanefsky R, Motamedi V, Mithani S, Mysliwiec V, Gill JM, Pattinson CL. Mild traumatic brain injuries with loss of consciousness are associated with increased inflammation and pain in military personnel. Psychiatry Res. 2019 Sep;279:34-39. doi: 10.1016/j.psychres.2019.07.001. Epub 2019 Jul 2. PMID 31280036
- [Result] Cairns BE, Arendt-Nielsen L, Sacerdote P. Perspectives in Pain Research 2014: Neuroinflammation and glial cell activation: The cause of transition from acute to chronic pain? Scand J Pain. 2015 Jan 1;6(1):3-6. doi: 10.1016/j.sjpain.2014.10.002. PMID 29911589
- [Result] Jodoin M, Rouleau DM, Gosselin N, Benoit B, Leduc S, Laflamme Y, Larson-Dupuis C, De Beaumont L. Comorbid mild traumatic brain injury increases pain symptoms in patients suffering from an isolated limb fracture. Injury. 2017 Sep;48(9):1927-1931. doi: 10.1016/j.injury.2017.06.025. Epub 2017 Jul 1. PMID 28693815
- [Result] Worden A, Ilyas AM. Ulnar neuropathy following distal humerus fracture fixation. Orthop Clin North Am. 2012 Oct;43(4):509-14. doi: 10.1016/j.ocl.2012.07.019. Epub 2012 Aug 30. PMID 23026466
- [Result] Mathew PK, Athwal GS, King GJ. Terrible triad injury of the elbow: current concepts. J Am Acad Orthop Surg. 2009 Mar;17(3):137-51. doi: 10.5435/00124635-200903000-00003. PMID 19264707
- [Result] Jodoin M, Rouleau DM, Charlebois-Plante C, Benoit B, Leduc S, Laflamme GY, Gosselin N, Larson-Dupuis C, De Beaumont L. Incidence rate of mild traumatic brain injury among patients who have suffered from an isolated limb fracture: Upper limb fracture patients are more at risk. Injury. 2016 Aug;47(8):1835-40. doi: 10.1016/j.injury.2016.05.036. Epub 2016 May 27. PMID 27291349
- [Result] Hansson E. Long-term pain, neuroinflammation and glial activation. Scand J Pain. 2010 Apr 1;1(2):67-72. doi: 10.1016/j.sjpain.2010.01.002. PMID 29913949
- [Result] Teunis T, Stoop N, Park CJ, Ring D. What factors are associated with a second opioid prescription after treatment of distal radius fractures with a volar locking plate? Hand (N Y). 2015 Dec;10(4):639-48. doi: 10.1007/s11552-015-9767-6. Epub 2015 Apr 30. PMID 26568716
- [Result] Butler MM, Ancona RM, Beauchamp GA, Yamin CK, Winstanley EL, Hart KW, Ruffner AH, Ryan SW, Ryan RJ, Lindsell CJ, Lyons MS. Emergency Department Prescription Opioids as an Initial Exposure Preceding Addiction. Ann Emerg Med. 2016 Aug;68(2):202-8. doi: 10.1016/j.annemergmed.2015.11.033. Epub 2016 Feb 11. PMID 26875061
- [Result] King NB, Fraser V, Boikos C, Richardson R, Harper S. Determinants of increased opioid-related mortality in the United States and Canada, 1990-2013: a systematic review. Am J Public Health. 2014 Aug;104(8):e32-42. doi: 10.2105/AJPH.2014.301966. Epub 2014 Jun 12. PMID 24922138
- [Result] Hina N, Fletcher D, Poindessous-Jazat F, Martinez V. Hyperalgesia induced by low-dose opioid treatment before orthopaedic surgery: An observational case-control study. Eur J Anaesthesiol. 2015 Apr;32(4):255-61. doi: 10.1097/EJA.0000000000000197. PMID 25485877
- [Result] Bot AG, Bekkers S, Arnstein PM, Smith RM, Ring D. Opioid use after fracture surgery correlates with pain intensity and satisfaction with pain relief. Clin Orthop Relat Res. 2014 Aug;472(8):2542-9. doi: 10.1007/s11999-014-3660-4. Epub 2014 Apr 29. PMID 24777731
- [Result] Glare P, Aubrey KR, Myles PS. Transition from acute to chronic pain after surgery. Lancet. 2019 Apr 13;393(10180):1537-1546. doi: 10.1016/S0140-6736(19)30352-6. PMID 30983589
- [Result] Grobet C, Marks M, Tecklenburg L, Audige L. Application and measurement properties of EQ-5D to measure quality of life in patients with upper extremity orthopaedic disorders: a systematic literature review. Arch Orthop Trauma Surg. 2018 Jul;138(7):953-961. doi: 10.1007/s00402-018-2933-x. Epub 2018 Apr 13. PMID 29654354
- [Result] de Putter CE, Selles RW, Polinder S, Panneman MJ, Hovius SE, van Beeck EF. Economic impact of hand and wrist injuries: health-care costs and productivity costs in a population-based study. J Bone Joint Surg Am. 2012 May 2;94(9):e56. doi: 10.2106/JBJS.K.00561. PMID 22552678
- [Result] Dietrich M, Wasmer M, Platz A, Spross C. Return-to-Work Following Open Reduction and Internal Fixation of Proximal Humerus Fractures. Open Orthop J. 2014 Sep 15;8:281-7. doi: 10.2174/1874325001408010281. eCollection 2014. PMID 25246994
- [Result] Fuzier R, Rousset J, Bataille B, Salces-y-Nedeo A, Magues JP. One half of patients reports persistent pain three months after orthopaedic surgery. Anaesth Crit Care Pain Med. 2015 Jun;34(3):159-64. doi: 10.1016/j.accpm.2014.09.006. Epub 2015 May 23. PMID 26004873
- [Result] Tunali O, Ersen A, Pehlivanoglu T, Bayram S, Atalar AC, Demirhan M. Evaluation of risk factors for stiffness after distal humerus plating. Int Orthop. 2018 Apr;42(4):921-926. doi: 10.1007/s00264-018-3792-3. Epub 2018 Feb 1. PMID 29392385